CLINICAL TRIAL: NCT00772668
Title: Pilot Study of RCVELP as First Line Therapy for Follicular Lymphoma (FL) and Marginal Zone Lymphoma (MZL)
Brief Title: Rituximab, Cyclophosphamide, Bortezomib, and Prednisone in Patients With Stage III/IV FL or MZL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Denise Pereira, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070963; SCCC-2006120 (Other: UM/Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2008-10-12; First posted 2008-10-15 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Bortezomib; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RCVELP (Experimental): Rituximab, Cyclophosphamide, Bortezomib, Prednisone (RCVELP):
  * Rituximab
    * Induction: 375 mg/m2 IV infusion on Day 1 of every 21 days cycle for 8 cycles
    * Maintenance: 375/m2 Days 1, 8, 15, 22 every 6 months for up to 4 cycles
  * Cyclophosphamide: 750 mg/m2 intravenous piggyback (IVPB) on Day 1 of every 21 day cycle for 8 cycles
  * Bortezomib: 1.6 mg/m2 IV push on Days 1 and 8 of every 21 days cycle for 8 cycles
  * Prednisone: 100 mg PO daily on Days 1-5 of every 21 day cycle for 8 cycles
  Interventions: Drug: Rituximab; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Administered intravenously during induction and maintenance therapy per protocol.
  Other Names: Rituxan
Drug: Bortezomib — Administered intravenously per protocol.
  Other Names: Velcade
Drug: Cyclophosphamide — Administered intravenously per protocol.
  Other Names: Cytoxan
Drug: Prednisone — Administered orally (PO) per protocol.
  Other Names: Deltasone

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving rituximab together with cyclophosphamide, bortezomib, and prednisone may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving rituximab together with cyclophosphamide, bortezomib, and prednisone works as first-line therapy in treating patients with stage III or stage IV follicular lymphoma or marginal zone lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

* Induction therapy: Patients receive rituximab IV and cyclophosphamide IV over 30 minutes on day 1, bortezomib IV on days 1 and 8, and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance therapy.
* Maintenance therapy: Patients receive rituximab IV on days 1, 8, 15, and 22. Treatment repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Histologically confirmed, untreated follicular lymphoma (FL) grade I, II or marginal zone lymphoma (MZL) Stage III or IV
* Presence of measurable or evaluable disease
* Age >17 years old
* Patients must have normal organ and marrow function as defined below, within 14 days of enrollment:

  * Serum bilirubin < 2.0 mg/dL
  * serum creatinine < 2 mg/dL unless due to lymphoma
  * Absolute Neutrophil Count (ANC) >1000/mm3
  * Platelets >100,000/mm3 unless due to lymphoma
  * Aspartate Transaminase (AST), Alanine Aminotransferase (ALT) and Alkaline phosphatase < 3x the upper limit of normal
* Eastern Cooperative Oncology Group (ECOG) performance status of 1, 2, 3
* No prior therapy for the FL or MZL including chemotherapy, single agent rituximab and radiation therapy
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria

* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 5), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient has hypersensitivity to boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* History of HIV infection (testing not required)
* Concurrent or previous malignancy whose prognosis is poor (< 90% probability of survival at 5 years) or those who are actively being treated for a second malignancy.

Ages: 17 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Pereira, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RCVELP
Started | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | RCVELP
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, According to the International Workshop Criteria (IWC) for Non-Hodgkin's Lymphoma (NHL)
Description: Rate of overall response (CR, CRu, PR) to protocol therapy according to International Workshop Criteria (IWC):
  * Complete Response (CR) includes complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities definitely assignable to NHL;
  * Complete Response Unconfirmed (CRu) includes above CR criteria but a residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the product of the perpendicular diameters (SPD), or indeterminate bone marrow;
  * Partial Response (PR) includes >= 50% decrease in SPD of the six largest dominant nodes or nodal masses, no increase in size of other nodes, liver or spleen.
Time Frame: Post cycles 2,4,6,8 and then every 3 months, about 2 years
Population: A minimum enrollment of 30 participants was required for this outcome measure. Due this minimum requirement not being met, and the early termination of the study due to lack of funding, the data for this outcome measure were not analyzed.
Arm/Group | RCVELP
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free-survival will be assessed according to according to the International Workshop Criteria (IWC). Progression-free survival will be measured as the time from date of enrollment to relapse, progression or death due to follicular lymphoma (FL) or marginal zone lymphoma (MZL), whichever occurs first. Participants who do not experience relapse or progression, and those who die from causes other than cancer, will be censored at the date of last contact.
Time Frame: Up to 5 years
Measure: Number; unit: months
Groups:
- RCVELP: Rituximab, Cyclophosphamide, Bortezomib, Prednisone (RCVELP):
  * Rituximab
    * Induction: 375 mg/m2 IV infusion on Day 1 of every 21 days cycle for 8 cycles
    * Maintenance: 375/m2 Days 1, 8, 15, 22 every 6 months for up to 4 cycles
  * Cyclophosphamide: 750 mg/m2 intravenous piggyback (IVPB) on Day 1 of every 21 day cycle for 8 cycles
  * Bortezomib: 1.6 mg/m2 IV push on Days 1 and 8 of every 21 days cycle for 8 cycles
  * Prednisone: 100 mg PO daily on Days 1-5 of every 21 day cycle for 8 cycles
  Rituximab: Administered intravenously during induction and maintenance therapy per protocol.
  Bortezomib: Administered intravenously per protocol.
  Cyclophosphamide: Administered intravenously per protocol.
  Prednisone: Administered orally (PO) per protocol.
Arm/Group | RCVELP
Number analyzed (Participants) | 3
months | NA — At the time of study termination, all participants were in remission. Progression Free Survival could not be measured as none of the participants progressed, and no mortality events have occurred.

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be measured as the time from date of enrollment to death from any cause. For patients who remain alive, survival time will be censored at the date of last contact.
Time Frame: Up to 5 years
Measure: Number; unit: months
Arm/Group | RCVELP
Number analyzed (Participants) | 3
months | NA — At the time of study termination, all participants were still alive. Overall Survival could not be measured as no mortality events have occurred.

4. Secondary Outcome: Rate of Toxicity in Study Participants
Description: Safety and tolerance to protocol therapy as evidenced by the rate of toxicity (serious adverse events and study-related adverse events) in study participants
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | RCVELP
Number analyzed (Participants) | 3
participants | 1

ADVERSE EVENTS:
Description: No non-serious study related adverse events were reported.
Arm/Group | RCVELP
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RCVELP (N=3)
Diverticulitis, Grade 3 (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of funding. All patients were removed from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes